CLINICAL TRIAL: NCT05991141
Title: Could Apnea Induce Hypoalgesia? An Explorative Randomized Controlled Trial
Brief Title: Could Apnea Induce Hypoalgesia?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Universitario La Salle (Other)
Responsible Party: Principal Investigator, José Fierro Marrero, Predoctoral researcher, Centro Universitario La Salle
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSEULS-PI-029/2022
Record Dates: First submitted 2023-07-26; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Pain; Apnea
Keywords: Pain; Apnoea; Apnea; Hypoalgesia
MeSH Terms: conditions — Pain; Apnea | interventions — N(6)-2-(4-aminophenyl)ethyladenosine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Experimental Group
  Interventions: Other: Apnea
- Control Group (Sham Comparator): Control Group
  Interventions: Other: Control Intervention

INTERVENTIONS:
Other: Apnea — In both experimental and control groups participants walked on a treadmill at 5.5 km/h with 5º inclination for 6 minutes. The experimental group (EG) added throughout the 6 minutes intervention the following breathing pattern cyclically: 5 seconds breathing normally followed by 10 seconds of low volume apnoea, performing a total of 24 cycles of normal breathing continued by apnoea.
  Arms: Experimental Group
Other: Control Intervention — In both experimental and control groups participants walked on a treadmill at 5.5 km/h with 5º inclination for 6 minutes. The Control group (CG) performed this protocol breathing normally.
  Arms: Control Group

SUMMARY:
A randomized controlled trial (RCT) in healthy subjects will be conducted with the following aims: (1) Explore the effect of low pulmonary volume dynamic apnoea bouts on Pressure Pain Threshold (PPT) and conditioned pain modulation (CPM); (2) analyse whether CPM response correlates with apnoea induced hypoalgesia; (3) examine the association between apnoea bouts, Rate of Perceived Exertion, hypoxemia and Heart Rate changes in PPT.

DETAILED DESCRIPTION:
A randomized controlled trial (RCT) in healthy subjects will be conducted with the following aims: (1) Explore the effect of low pulmonary volume dynamic apnoea bouts on Pressure Pain Threshold (PPT) and conditioned pain modulation (CPM); (2) analyse whether CPM response correlates with apnoea induced hypoalgesia; (3) examine the association between apnoea bouts Rate of Perceived Exertion, hypoxemia and Heart Rate changes in PPT

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants
* 18-30 years
* Currently pain-free
* Basal SpO2 ≥95%

Exclusion Criteria:

* Diabetes diagnosis
* Hypertension or hypotension diagnosis
* Pharmacological treatment
* Frequent pain during last month
* Drug consumption
* Self-harming behaviours
* Pregnant or potentially pregnant
* Cardiac or respiratory pathology
* Splenectomy or spleen disease
* Having performed moderate or high intensity physical activity 24 hours prior to the study
* Not having slept the previous night
* Alcohol intake 24 hours prior to study.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Pressure Pain Threshold | Before and immediately after the interventions
  PPT refers to the minimal amount of pressure needed to cause the first sensation of pain. The mechanical pressure algometer (PAIN TEST™ FPX 25, Wagner Instruments, Greenwich, CT, USA) counted with a round rubber disc of 1 cm2, displaying values in Kg, hence, data was expressed in Kg/cm2. Two locations, in upper and lower limbs, were examined to examine systemic hypoalgesia effects. The dorsal distal-phalange base of the thumb and tibialis anterior muscle belly, both in the dominant limb, were tested. These regions were marked with a pen before assessments, to repeat the trials in the same place. Three trials were tested in each location, with 30 seconds rest between trials. Pressure speed was paced with a metronome applying a constant force of 0.5 Kg/cm2/s ± 0.1 Kg/cm2/s.

SECONDARY OUTCOMES:
Conditioned pain modulation | Before and immediately after the interventions
  Conditioning stimulus was applied on the contralateral limb to test stimulus, since its arrangement does not influence CPM response. Only controversial CPM response have appeared when tests and conditioned stimuli were applied on the same body region. Ischemic pain was applied as conditioning stimulus and PPT as test stimulus. Ischemic pain was provoked inflating a sphygmomanometer at the proximal region of the non-dominant arm. When inflated up to 180-200 mmHg patients were asked to actively move fingers and wrist. They were asketd to report when a 7/10 pain in Numerical Pain Rating Scale (NPRS) scale was reached. In that moment, three trials of test stimuli were applied on the dorsal distal-phalange base of the thumb in the dominant arm, while maintaining the ischemic pain perception.
Heart Rate and Oxygen Saturation | During the intervention and for 2 minutes additionally after the end of the intervention
  We video-taped HR and SpO2 values during the 6 min interventions and 2 minutes afterwards to explore their changes during and after interventions. HR and SpO2 data were extracted in each second. These values would be graphically displayed. Peak %HRmax and minimum SpO2, and means of both variables, value would be extracted from the 6-minute interventions. HR zones or exercise-induced hypoxemia zones were also recorded.
Rated Perceived Exertion | This outcome was assessed immediately after having finished the intervention protocols
  Apnea and control interventions were explored in terms of Rated Perceived Exertion in with Borg's modified CR-10

CONTACTS AND LOCATIONS:
Overall Officials: José Fierro Marrero, Principal Investigator — CSEULaSalle
Locations (1):
- Centro Superior de Estudios La Salle, Madrid, Spain

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-02-27): https://cdn.clinicaltrials.gov/large-docs/41/NCT05991141/SAP_000.pdf